CLINICAL TRIAL: NCT05283044
Title: Implementing Precision Medicine in cOmmunity HospiTALs
Acronym: PRISM-POrTAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-A02862-39; 2021/3331 (Other: CSET number)
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Liquid Biopsy

STUDY DESIGN:
Intervention Model Description: Proportion of patients presenting for whom ct DNA sequencing has allowed to propose a systemic treatment that was not considered before by the clinician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biopsy liquid contributive (Other): Patients presenting for whom ct DNA sequencing
  Interventions: Biological: biopsy liquid

INTERVENTIONS:
Biological: biopsy liquid — Patient performs a blood test at treatment baseline

SUMMARY:
This is a prospective biomarker study that aims at demonstrating the impact of liquid biopsy to deliver better treatment for cancer patients with metastatic disease managed in the community setting

DETAILED DESCRIPTION:
Patients will be selected to present a metastatic cancer (de novo or relapse after primary tumor treatment) eligible for a first line treatment (chemotherapy, immunotherapy, endocrine therapy or targeted therapy).

All tumor subtype could be enrolled in the study; metastatic prostate cancer must be resistant to castration. Triple negative breast cancer and Hormone receptor positive, Her2-negative metastatic breast cancer resistant to endocrine therapy are eligible to the study.

A plasma sample will be collected at baseline and will be tested for a large panel of gene and MSI status using Next Generation Sequencing (NGS) (cf table). Results will be discussed within a Molecular Tumor Board (MTB) with all declared centers.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if they meet all of the following criteria:

1. Age ≥ 18 years
2. Histology: solid malignant tumor
3. Locally advanced/unresectable and/or metastatic (for prostate cancer: castration resistant prostate cancer, for RH+/HER2- breast cancer: prior treatment with endocrine therapy plus anti-CDK4/6 inhibitor)
4. Eastern Cooperative Oncology Group (ECOG) performance status < 2
5. Measurable disease as per RECIST criteria
6. Patient with a social security in compliance with the French law relating to biomedical research (Article L.1121-11 of French Public Health Code)
7. Voluntary signed and dated written informed consent prior to any study specific procedure.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Radiological evidence of symptomatic or progressive brain metastases
2. Previous or current malignancies of others histologies within the last 2 years, with the exception of in situ carcinoma of the cervix, and adequately treated basal cell or squamous cell carcinoma of the skin and prostate cancer
3. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in a clinical trial or which would jeopardize compliance with the protocol
4. Patient under guardianship or deprived of his liberty by a judicial or administrative decision or incapable of giving its consent
5. Minors (Age < 18 years)
6. Pregnant or breast-feeding women
7. Previous enrollment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2028-11-15 (Estimated); Study Completion 2030-04-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients for whom ctDNA sequencing | 72 months
  The primary objective of the study will be to evaluate the impact of ctDNA sequencing on the treatment plan of cancer patients managed in satellite centers. This will be performed by estimating the proportion of patients for whom ctDNA sequencing has allowed to propose a systemic treatment that was not considered before the clinician.

SECONDARY OUTCOMES:
Utilization rates of molecular profiling information | 72 months
  The utilization rates of molecular profiling information (including utilization of information for standard regimens or clinical trials of molecularly targeted therapies)
Rate of molecular screening failure | 72 months
Relapsed time between liquid biopsy and matched therapy onset | 72 months
Rate of patients presenting targetable alterations | 72 months
  The rate of patients presenting targetable alterations according to alterations subtypes (copy number/mutation/oncogenic fusions)
Utilization rate of tumor mutational burden | 72 months
  The utilization rate of tumor mutational burden (TMB - based on new generation sequencing panels)
Objective Response Rate | 72 months
Overall Survival of patients treated with a therapy matched to a targetable alteration and recommended by the MTB based on the ctDNA sequencing | 72 months

CONTACTS AND LOCATIONS:
Locations (21):
- France (19):
  - CH de la Côte Basque, Bayonne
  - CH de Bligny, Bligny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH Sud Francilien, Corbeil-Essonnes
  - CH Annecy Genevois, Épagny
  - GHM de Grenoble, Grenoble
  - CHU de La Réunion, La Réunion
  - Clinique Saint-Jean l'ermitage, Melun
  - Hôpital Américain, Neuilly-sur-Seine
  - Hôpital de la source - CHR d'Orléans, Orléans
  - Hôpital Saint-Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Groupement Hospitalier Diaconesses-Croix, Paris
  - Centre Hospitalier, Pau
  - Centre Eugène Marquis, Rennes
  - Hôpitaux Privés de la Loire, Saint-Etienne
  - HIA Bégin, Saint-Mandé
  - Hôpital Foch, Suresnes
  - Hôpital Nord-Ouest Villefranche-sur-Saône, Villefranche-sur-Saône
- CHPF, Pirae, French Polynesia
- Clinique Kuindo Magnin, Noumea, New Caledonia

IPD SHARING:
Plan to Share IPD: No
no IPD in this study